CLINICAL TRIAL: NCT05373628
Title: Quantitative Parameters of Cell Size Imaging: Correlation With Histopathological Features in Patients With Breast Cancer
Brief Title: Study on the Correlation Between the Quantitative Parameters of Mr Mean Cell Size Imaging and the Histopathological Characteristics of Breast Cancer
Acronym: OGSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiang Zhang, Department of Radiology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSEC-KY-KS-2022-056
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Breast Carcinoma; Magnetic Resonance Imaging；OGSE
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gradient and pulse imaging (Experimental): All subjects used standardized breast MRI scanning schemes, including T2 weighted imaging (T2WI), T1 weighted imaging (T1WI), diffusion weighted imaging (DWI), PGSE, OGSE and contrast dynamic enhancement (DCE). Three quantitative parameters of VIN, DEX and D are derived on MATLAB software
  Interventions: Diagnostic Test: Gradient and pulse imaging

INTERVENTIONS:
Diagnostic Test: Gradient and pulse imaging — A novel diffusion-based magnetic resonance imaging method

SUMMARY:
Patients with breast masses and suspected breast malignancies by ultrasound / mammography were prospectively included. After routine MRI scanning, all patients underwent average cell size imaging sequence scanning, and finally underwent breast MRI enhanced scanning. Inclusion criteria of breast cancer patients: (1) breast cancer confirmed by surgery or biopsy; (2) The status of estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor-2 (HER-2), Ki-67 and lymphatic vessel invasion (LVI) in breast cancer were clearly diagnosed by pathology; (3) Routine MRI, PGSE and OGSE scans were performed within 1 week before pathological examination. Exclusion criteria: (1) breast tumor patients who had received treatment before PGSE and OGSE sequence scanning; (2) Patients who underwent breast tumor puncture within 2 weeks before PGSE and OGSE sequence scanning; (3) Patients with breast masses without surgery or biopsy after PGSE and OGSE sequence scanning; (4) The breast mass was confirmed to be other diseases except breast cancer by pathological examination; (5) Due to poor image quality caused by motion artifacts or other reasons, PGSE and OGSE sequence post-processing cannot be carried out. All subjects were required to sign written informed consent.

Breast MRI data were collected using Philips ingenia DNA 3T MR scanner in the Netherlands. All subjects used standardized breast MRI scanning schemes, including T2 weighted imaging (T2WI), T1 weighted imaging (T1WI), diffusion weighted imaging (DWI), PGSE, OGSE and contrast dynamic enhancement (DCE). Three quantitative parameters of VIN, DEX and D were derived from MATLAB software. The correlation between the quantitative parameters of mean cell size imaging and pathological indexes Er, PR, HER-2, Ki-67 and LVI was evaluated by Spearman correlation analysis. The predictive factors of the quantitative parameters of mean cell size model for different pathological characteristics of breast cancer were determined by logistic regression model, The diagnostic efficacy of quantitative parameters of mean cell size model for pathological classification indexes was evaluated by subject operating characteristic (ROC) curve and area under curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer was confirmed by operation or biopsy;
2. The status of estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor-2 (HER-2), Ki-67 and lymphatic vessel invasion (LVI) in breast cancer were clearly diagnosed by pathology;
3. Routine MRI and mean cell size imaging sequence scanning were performed within 1 week before pathological examination

Exclusion Criteria:

(1) Breast cancer patients who had received treatment before mean cell size imaging sequence scanning; (2) Patients who had undergone breast tumor puncture within 2 weeks before the mean cell size imaging sequence scan; (3) Patients with breast masses without surgery or biopsy after mean cell size imaging sequence scanning; (4) The breast mass was confirmed to be other diseases except breast cancer by pathological examination; (5) The image quality is poor due to motion artifacts or other reasons, so the average cell size imaging post-processing cannot be carried out.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-11 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic characteristic | Up to 2 months
  Estrogen receptor (ER) status of breast cancer
2. Pathologic characteristic | Up to 2 months
  Progesterone receptor (PR) status of breast cancer

OTHER OUTCOMES:
Pathologic characteristic | Up to 2 months
  Human epidermal growth factor 2 (HER-2) status of breast cancer
Pathologic characteristic | Up to 2 months
  Ki-67 status of breast cancer
Pathologic characteristic | Up to 2 months
  Lymphatic vessel invasion (LVI) status of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xiang, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiology, Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Su Y, Qiu Y, Huang X, Peng Y, Yang Z, Ding M, Hu L, Wang Y, Zhao C, Qian W, Zhang X, Shen J. Benign and Malignant Breast Lesions: Differentiation Using Microstructural Metrics Derived from Time-Dependent Diffusion MRI. Radiol Imaging Cancer. 2025 May;7(3):e240287. doi: 10.1148/rycan.240287. PMID 40214515